CLINICAL TRIAL: NCT01400334
Title: Hibernating Myocardium and Sudden Cardiac Death
Brief Title: Prediction of ARrhythmic Events With Positron Emission Tomography
Acronym: PAREPET
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, JOHN CANTY, Principal Investigator, State University of New York at Buffalo
Other Study IDs: HL76252
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Ischemic Cardiomyopathy; Hibernating Myocardium; Nerve; Disorder, Sympathetic
Keywords: Ischemic Cardiomyopathy; Sudden Cardiac Death; Positron Emission Tomography; Hibernating Myocardium; Denervated Myocardium
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ischemic Cardiomyopathy: Subjects with ischemic cardiomyopathy [pre-enrollment left ventricular ejection fraction ≤0.35, with coronary artery disease documented by cardiac catheterization, a history of definite myocardial infarction, or reversible ischemia on nuclear imaging] who are considered eligible to receive an implantable cardiac defibrillator for the primary prevention of sudden cardiac death.
  Interventions: Radiation: Positron Emission Tomography

INTERVENTIONS:
Radiation: Positron Emission Tomography — Quantification of cardiac function using positron emission tomography and: a)11C-meta-hydroxyephedrine [HED, 20 mCi (740 MBq)] to quantify sympathetic nerve function, b) 13N-ammonia [NH3, 20 mCi (740 MBq)] for regional perfusion, and c) 18F-2-deoxyglucose [FDG; 6.5 mCi (241 MBq)] administered during a hyperinsulinemic-euglycemic clamp to assess viability.

SUMMARY:
The hypothesis of PAREPET is that hibernating myocardium (viable myocardium with reduced resting flow) and/or viable but denervated myocardium can predict the risk of sudden death in subjects with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Currently available electrophysiological approaches are limited in their ability to identify the majority of patients with CAD and LV dysfunction that succumb to sudden cardiac death (SCD). Half of the patients developing SCD are not inducible at electrophysiological testing underscoring the need for new ways to identify substrates leading to arrhythmic death. Viable chronically dysfunctional with reduced resting flow, or hibernating myocardium, not amenable to revascularization appears to be a major risk factor for subsequent cardiac death and is present in up to 60% of patients with ischemic cardiomyopathy. Cause specific mortality data is limited but appears to be arrhythmic rather than from fatal myocardial infarction or progressive heart failure. Revascularization improves survival but most patients with hibernating myocardium are managed medically due to prohibitive procedural risks or technical limitations. Basic studies in swine with hibernating myocardium demonstrate SCD arising from VT/VF in the absence of myocardial scar or heart failure. The central hypothesis of this proposal is that the presence of hibernating myocardium as opposed to scar identifies a large subset of patients with ischemic cardiomyopathy that are at high risk for SCD. We further hypothesize that this risk is related to inhomogeneity in sympathetic innervation arising from chronic repetitive ischemia. PAREPET is a prospective observational study that will enroll patients with coronary disease, Class I-III heart failure and an ejection fraction ≤35%. Using positron emission tomography (PET), the frequency and amount of hibernating myocardium will be quantified in patients that are not candidates for coronary revascularization. Three Specific Aims are proposed. Aim 1 will determine whether imaging the mismatch between viability (preserved 18F-2-deoxyglucose) and reduced resting flow (13NH3) can predict an increased risk of SCD (or ICD discharge for VT/VF as a surrogate end-point) in hibernating myocardium. Aim 2 will image norepinephrine uptake using 11C-hydroxyephedrine to determine whether inhomogeneity in myocardial sympathetic innervation predicts SCD risk better than viability testing. Aim 3 will identify whether the substrate identified by PET is stable after an aborted SCD event by evaluating temporal changes in function, viability and sympathetic innervation in patients with an ICD. Our long-term objective is to develop better approaches to identify patients with CAD who are most likely to benefit from primary prevention of SCD with placement an ICD.

ELIGIBILITY:
Inclusion Criteria:

* LV EF ≤35% (by nuclear imaging, cardiac catheterization or echocardiography)
* Coronary artery disease documented by cardiac catheterization, a history of definite myocardial infarction, or reversible ischemia on nuclear imaging
* New York State Heart Association functional Class I-III heart failure
* Not a candidate for surgical or percutaneous coronary revascularization at the time of enrollment

Exclusion Criteria:

* History of resuscitated sudden cardiac death, sustained ventricular tachycardia, appropriate implantable cardiac defibrillator (ICD) discharge, or unexplained syncope
* Myocardial infarction within 30 days
* Coronary artery bypass grafting within 1 year
* Percutaneous intervention within 3 months
* Claustrophobia or physical limitation that would preclude PET scanning
* Pregnancy
* Tricyclic antidepressant drug therapy
* Comorbidities that would be expected to result in noncardiac death within 2 years
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Western New York referred for an implantable cardiac defibrillator, transthoracic echocardiography, and/or coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2004-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sudden Cardiac Death | every 3 months
  Adjudicated sudden cardiac death and implantable cardiac defibrillator therapy for fast ventricular tachycardia (>240 bpm) or ventricular fibrillation.

SECONDARY OUTCOMES:
Cardiac Death | every 3 months
  Sudden cardiac death and adjudicated non-sudden cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: John M Canty, MD, Principal Investigator — State University of New York at Buffalo; James A Fallavollita, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- SUNYBuffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Fallavollita JA, Luisi AJ Jr, Michalek SM, Valverde AM, deKemp RA, Haka MS, Hutson AD, Canty JM Jr. Prediction of arrhythmic events with positron emission tomography: PAREPET study design and methods. Contemp Clin Trials. 2006 Aug;27(4):374-88. doi: 10.1016/j.cct.2006.03.005. Epub 2006 May 2. PMID 16647885
- [Result] Fallavollita JA, Heavey BM, Luisi AJ Jr, Michalek SM, Baldwa S, Mashtare TL Jr, Hutson AD, Dekemp RA, Haka MS, Sajjad M, Cimato TR, Curtis AB, Cain ME, Canty JM Jr. Regional myocardial sympathetic denervation predicts the risk of sudden cardiac arrest in ischemic cardiomyopathy. J Am Coll Cardiol. 2014 Jan 21;63(2):141-9. doi: 10.1016/j.jacc.2013.07.096. Epub 2013 Sep 25. PMID 24076296
- [Result] Al-Zaiti SS, Fallavollita JA, Canty JM Jr, Carey MG. Electrocardiographic predictors of sudden and non-sudden cardiac death in patients with ischemic cardiomyopathy. Heart Lung. 2014 Nov-Dec;43(6):527-33. doi: 10.1016/j.hrtlng.2014.05.008. Epub 2014 Jul 2. PMID 24996250
- [Result] Al-Zaiti SS, Fallavollita JA, Wu YW, Tomita MR, Carey MG. Electrocardiogram-based predictors of clinical outcomes: a meta-analysis of the prognostic value of ventricular repolarization. Heart Lung. 2014 Nov-Dec;43(6):516-26. doi: 10.1016/j.hrtlng.2014.05.004. Epub 2014 Jun 29. PMID 24988910
- [Derived] Zelt JGE, Wang JZ, Mielniczuk LM, Beanlands RSB, Fallavollita JA, Canty JM Jr, deKemp RA. Positron Emission Tomography Imaging of Regional Versus Global Myocardial Sympathetic Activity to Improve Risk Stratification in Patients With Ischemic Cardiomyopathy. Circ Cardiovasc Imaging. 2021 Jun;14(6):e012549. doi: 10.1161/CIRCIMAGING.121.012549. Epub 2021 Jun 9. PMID 34102857
- [Derived] Fallavollita JA, Dare JD, Carter RL, Baldwa S, Canty JM Jr. Denervated Myocardium Is Preferentially Associated With Sudden Cardiac Arrest in Ischemic Cardiomyopathy: A Pilot Competing Risks Analysis of Cause-Specific Mortality. Circ Cardiovasc Imaging. 2017 Aug;10(8):e006446. doi: 10.1161/CIRCIMAGING.117.006446. PMID 28794139
- [Derived] Cain ME. Impact of denervated myocardium on improving risk stratification for sudden cardiac death. Trans Am Clin Climatol Assoc. 2014;125:141-53; discussion 153. PMID 25125727